CLINICAL TRIAL: NCT01034059
Title: Assessment of sTREM-1 as a Diagnostic Marker in Patients With Neutropenic Fever
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Szu-Chun Hsu, Department of Laboratory Medicine, National Taiwan University Hospital and College of Medicine, Taipei
Other Study IDs: 200806051R
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Neutropenic Fever
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The soluble triggering receptor expressed on myeloid cells-1 (sTREM-1) was an established biomarker useful for infection in non-neutropenic patients. In this study, we tested sTREM-1 in the patients with neutropenic fever. Pro-calcitonin (PCT) and C-reactive protein (CRP) were also measured. We planned to investigate and explore the role of sTREM-1 in early diagnosis of infection in patients with neutropenic fever.

DETAILED DESCRIPTION:
Patients with hematological malignancies developed neutropenia after chemotherapy. We checked the serum level of sTREM-1 in patients with neutropenic fever. Those patients were classified to 2 groups: documented infection or low likelihood of infection. Their sTREM-1 level was measured and was compared with other biomarker such as CRP and procalcitonin. The value of sTREM-1 for diagnosis of infection in patients with neutropenic fever was thus evaluated.

ELIGIBILITY:
Inclusion Criteria:

* chemotherapy-related neutropenia (granulocytes < 0.5 × 109/l or leukocytes < 1 × 109/l) and fever (body temperature > 38.0°C over a 6 hour observation period or body temperature ≥ 38.5°C once.

Exclusion Criteria:

* prolonged fever before presenting for admission,
* antibiotics therapy in the past 72 hours,
* more than two sites of infectious focus,
* concomitant solid organ malignancy and blast in hemogram.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hematological malignancy developing neutropenic fever after chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Chun Hsu, MD, Principal Investigator — Department of Laboratory Medicine, National Taiwan University Hospital and College of Medicine, Taipei